CLINICAL TRIAL: NCT01144299
Title: A Phase III Study for Evaluation of Immunogenicity and Reactogenicity of Fluarix™/Influsplit SSW® 2010/2011 in People Aged 18 Years or Above
Brief Title: A Study to Evaluate the Safety and Immunogenicity of GSK Biologicals' Seasonal Influenza Vaccine in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 114292
Record Dates: First submitted 2010-06-10; First posted 2010-06-15 (Estimated); Results first posted 2010-10-27 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2016-09

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human

ARMS (2):
- Fluarix Adult Group (Experimental): Subjects aged 18 to 60 years received one dose of Fluarix™.
  Interventions: Biological: Fluarix™/Influsplit SSW®
- Fluarix Elderly Group (Experimental): Subjects aged > 60 years received one dose of Fluarix™.
  Interventions: Biological: Fluarix™/Influsplit SSW®

INTERVENTIONS:
Biological: Fluarix™/Influsplit SSW® — Single intramuscular dose on Day 0

SUMMARY:
This study is designed to test the immunogenicity and reactogenicity of the Fluarix™/Influsplit SSW® influenza vaccine containing the influenza strains recommended for the 2010-2011 season.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female aged 18 years or above at the time of the vaccination.
* Written informed consent obtained from the subject.
* Healthy subjects or with well-controlled chronic diseases as established by medical history and clinical examination before entering into the study.
* If the subject is female, she must be of non-childbearing potential or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the vaccination or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the vaccine dose.
* Administration of immunoglobulins and/or any blood products within the three months preceding the administration of the study vaccine or planned during the study.
* Administration of an influenza vaccine within 6 months preceding the study start.
* Administration of an influenza vaccine other than the study vaccine during the entire study
* Clinically or virologically confirmed influenza infection within 6 months preceding the study start
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute disease at the time of enrolment.
* Acute clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Not stabilized or clinically serious chronic underlying disease.
* Lactating female.
* History of chronic alcohol consumption and/or drug abuse.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Any condition which, in the opinion of the investigator, prevents the subject from participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2010-06-17; Primary Completion 2010-07-10 (Actual); Study Completion 2010-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Germany (2):
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Freital, Saxony

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 114292 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114292 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114292 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114292 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114292 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114292 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114292 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluarix Adult Group | Fluarix Elderly Group
Started | 60 | 54
Completed | 58 | 54
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluarix Adult Group | Fluarix Elderly Group | Total
Number analyzed (Participants) | 60 | 54 | 114
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.1 (13.10) | 68.6 (5.08) | 52.1 (18.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 26 | 58
  Male | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Hemagglutination Inhibition (HI) Antibody Titer
Description: Titers given as geometric mean titer (GMT) were presented for all three vaccine influenza virus strains
Time Frame: Day 0 and Day 21
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for analysis of immunogenicity, on subjects with available data
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Fluarix Adult Group | Fluarix Elderly Group
Number analyzed (Participants) | 55 | 53
titer
  A/California (Day 0) | 10.2 [7.7 to 13.6] | 8.7 [6.6 to 11.4]
  A/California (Day 21) | 314.1 [237.5 to 415.4] | 89.4 [60.1 to 133.0]
  A/Victoria (Day 0) | 15.2 [11.6 to 20.0] | 10.5 [8.3 to 13.3]
  A/Victoria (Day 21) | 89.6 [70.8 to 113.3] | 75.4 [56.8 to 100.2]
  B/Brisbane (Day 0) | 36.3 [26.4 to 50.1] | 42.1 [30.6 to 57.9]
  B/Brisbane (Day 21) | 271.6 [213.3 to 345.9] | 132.3 [99.0 to 176.9]

2. Primary Outcome: Number of Seroprotected Subjects
Description: A seroprotected subject is a subject with a serum HI antibody titer ≥ 1:40
Time Frame: Day 0 and Day 21
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, on subjects with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Adult Group | Fluarix Elderly Group
Number analyzed (Participants) | 55 | 53
Participants
  A/California (Day 0) | 9 | 4
  A/California (Day 21) | 54 | 41
  A/Victoria (Day 0) | 14 | 7
  A/Victoria (Day 21) | 48 | 45
  B/Brisbane (Day 0) | 29 | 29
  B/Brisbane (Day 21) | 55 | 47

3. Primary Outcome: Number of Seroconverted Subjects
Description: A seroconverted subject is a subject with a pre-vaccination serum HI titer < 1:10 and a post-vaccination serum HI titer ≥ 1:40, or a pre-vaccination serum HI titer ≥ 1:10 and a fold increase (Day 21/Day 0) ≥ 4
Time Frame: Day 21
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, on subjects with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Adult Group | Fluarix Elderly Group
Number analyzed (Participants) | 55 | 53
Participants
  A/California | 50 | 35
  A/Victoria | 35 | 36
  B/Brisbane | 33 | 18

4. Primary Outcome: Seroconversion Factor
Description: Seroconversion factor, defined as the fold increase in serum HI GMT post-vaccination compared to pre-vaccination (Day 0), is presented for all three vaccine influenza virus strains
Time Frame: Day 21
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, on subjects with available data
Measure: Mean (95% Confidence Interval); unit: fold change
Arm/Group | Fluarix Adult Group | Fluarix Elderly Group
Number analyzed (Participants) | 55 | 53
fold change
  A/California | 30.8 [21.8 to 43.5] | 10.3 [7.0 to 15.2]
  A/Victoria | 5.9 [4.5 to 7.8] | 7.2 [5.1 to 10.1]
  B/Brisbane | 7.5 [5.1 to 11.0] | 3.1 [2.2 to 4.4]

5. Primary Outcome: Seroprotection Power
Description: Seroprotection power is defined as the number of subject who had a pre-vaccination titer < 1:40 and a post-vaccination titer ≥ 1:40
Time Frame: Day 21
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity, on subjects with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Adult Group | Fluarix Elderly Group
Number analyzed (Participants) | 46 | 49
Participants
  A/California | 45 | 37
  A/Victoria: number analyzed (Participants) | 41 | 46
  A/Victoria | 34 | 38
  B/Brisbane: number analyzed (Participants) | 26 | 24
  B/Brisbane | 26 | 18

6. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed include ecchymosis, induration, pain, redness, and swelling.
Time Frame: During the 4-day (Day 0-3) post-vaccination period
Population: Analysis was performed on the Total Vaccinated Cohort, on subjects with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Adult Group | Fluarix Elderly Group
Number analyzed (Participants) | 59 | 54
Participants
  Ecchymosis | 3 | 0
  Induration | 9 | 9
  Pain | 40 | 17
  Redness | 10 | 15
  Swelling | 8 | 7

7. Secondary Outcome: Number of Subjects Reporting Solicited General Symptoms
Description: Solicited general symptoms assessed include arthralgia, fatigue, headache, myalgia, shivering, sweating, and fever.
Time Frame: During the 4-day (Day 0-3) post-vaccination period
Population: Analysis was performed on the Total Vaccinated Cohort, on subjects with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Adult Group | Fluarix Elderly Group
Number analyzed (Participants) | 59 | 54
Participants
  Arthralgia | 6 | 4
  Fatigue | 13 | 8
  Headache | 11 | 9
  Myalgia | 11 | 9
  Shivering | 5 | 3
  Fever (Axillary) | 1 | 0
  Sweating | 3 | 3

8. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AE)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product
Time Frame: During the 21-day (Day 0-20) post-vaccination period
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Adult Group | Fluarix Elderly Group
Number analyzed (Participants) | 60 | 54
Participants | 12 | 6

9. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAE)
Description: An SAE is any untoward medical occurrence that: results in death, is lifethreatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: During the entire study period (From Day 0 up to Day 21)
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Adult Group | Fluarix Elderly Group
Number analyzed (Participants) | 60 | 54
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Fluarix Adult Group | Fluarix Elderly Group
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/54
Other Adverse Events (participants affected / at risk) | 50/60 | 30/54
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluarix Adult Group (N=60) | Fluarix Elderly Group (N=54)
Ecchymosis (General disorders) | 3 | 0
Induration (General disorders) | 9 | 9
Pain (General disorders) | 40 | 17
Redness (General disorders) | 10 | 15
Swelling (General disorders) | 8 | 7
Arthralgia (General disorders) | 6 | 4
Fatigue (General disorders) | 13 | 8
Headache (General disorders) | 11 | 9
Myalgia (General disorders) | 11 | 9
Shivering (General disorders) | 5 | 3
Sweating (General disorders) | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.